CLINICAL TRIAL: NCT04685655
Title: RescuE pLAsma eXchange in Severe COVID-19 (RELAX Severe COVID-19)
Brief Title: RescuE pLAsma eXchange in Severe COVID-19
Acronym: RELAX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low numbers of severe COVID-19 cases with current variants.
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Christian Nusshag, MD, Attending, Department of Nephrology, University Hospital Heidelberg
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-911/2020
Record Dates: First submitted 2020-12-23; First posted 2020-12-28 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Therapeutic Plasma Exchange; Covid19
Keywords: Plasma exchange; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Plasma Exchange

STUDY DESIGN:
Intervention Model Description: Therapeutic plasma exchange in patients with severe COVID 19
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 therapy according to center standard alone (No Intervention)
- Therapeutic plasma exchange and COVID-19 therapy according to center standard (Active Comparator)
  Interventions: Other: Therapeutic plasma exchange

INTERVENTIONS:
Other: Therapeutic plasma exchange — Treatment with therapeutic plasma exchange. Plasma from healthy donors is used.
  Arms: Therapeutic plasma exchange and COVID-19 therapy according to center standard

SUMMARY:
The spectrum of coronavirus disease 2019 (COVID-19) ranges from asymptomatic infection to acute respiratory distress syndrome ("ARDS") and patient death. Severely affected patients may develop a cytokine storm-like clinical syndrome with high mortality. Laboratory tests in these patients show an excessive and uncontrolled immune response with consecutive multi-organ failure. In addition, there is evidence for the development of prothrombotic autoantibodies as an epiphenomenon of "Severe Acute Respiratory Syndrome Coronavirus 2" (SARS-CoV-2) infection. Therapeutic plasma exchange ("TPE") is being discussed as a therapeutic alternative in patients with severe, refractory COVID-19. The idea is that plasma exchange eliminates both endogenous and exogenous inducers of an exuberant inflammatory response as well as prothrombotic factors, thus breaking the secondary vicious circle of SARS-CoV-2 infection. In general, TPE is a safe procedure with known efficacy in other severe viral diseases as well as in cytokine storm-like diseases and ARDS of other geneses. Moreover, initial data, mostly derived from case studies, demonstrate promising therapeutic efficacy of TPE in severe COVID-19 courses with previously lacking treatment options. To further evaluate the therapeutic efficacy of TPE in severe COVID-19, a prospective randomized controlled trial of TPE in severe SARS-CoV-2 infection is being conducted at our center. Patients will be randomized to a control group (standard therapy according to center standards) and a therapy/intervention group (standard therapy + TPE).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by the study participant or their legally appointed representative.
* Age ≥ 18 years
* Evidence of acute SARS-CoV-2 infection, confirmed by PCR testing
* Invasive ventilation
* Fever ≥ 38.5°C, confirmed by a total of 3 consecutive measurements or ongoing renal replacement therapy and temperature ≥ 37.5°C
* D-dimers ≥ 2mg/L
* Dexamethasone ≥ 6mg/day or equivalent dose on at least 2 days

Exclusion Criteria:

* Age > 85 years
* Pre-existing treatment limitations
* Pregnancy
* Confirmed pulmonary arterial embolism with hemodynamically relevant right heart strain
* ST-segment elevation myocardial infarction (STEMI)
* Participation in an intervention study elsewhere

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Survival | 30 days after randomization
  Intention to treat analysis

SECONDARY OUTCOMES:
Survival | 15, 30, 60, 90, 365 days after randomization
  Intention to treat & per protocol
Ventilator-free days | 15, 30, 60, 90 days after randomization
Length of hospital an ICU stay | through study completion, an average of 1 year
Improvement defined as two points on seven point ordinal WHO scale | through study completion, an average of 1 year
Reduction of vasopressors after TPE treatments | through study completion, an average of 1 year
Incidence of acute kidney injury, renal replacement therapy and renal recovery | 15, 30, 60, 90 days after randomization
  AKI KDIGO criteria
Frequency of typical complications associated to therapeutic plasma exchange | through study completion, an average of 1 year
Reduction of inflammation mediators, (auto-)antibodies, and coagulation-associated molecules and their temporal correlation to TPE | through study completion, an average of 1 year
D-dimer-dependent assessment of therapeutic efficacy. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Heidelberg University Hospital, Heidelberg, Baden-Wurttemberg
  - Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg
  - University Hospital Essen, Essen, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Undecided
On request